CLINICAL TRIAL: NCT02097316
Title: Feasibility Study of the JewelPump Version 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A00792-43
Record Dates: First submitted 2013-09-26; First posted 2014-03-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes
Keywords: Glycemic control; JewelPump accuracy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- JewelPump (Experimental): JewelPump for the first treatment period followed by the usual pump for the second treatment period
  Interventions: Device: JewelPump; Device: usual insulin pump
- Usual insulin pump (Active Comparator): Patients in the arm 2, will have the usual insulin pump for the first treatment period, followed with the second period which they will have the JewelPump.
  Interventions: Device: JewelPump; Device: usual insulin pump

INTERVENTIONS:
Device: JewelPump
Device: usual insulin pump

SUMMARY:
The study will be conducted, in cross-over with a time interval of at least 2 days between 2 treatment periods. Patients will be randomized into 2 groups According to the order of the randomization, patients will bear the JewelPump for 5 days, followed by a period of 5 days of treatment with their usual pumps.

DETAILED DESCRIPTION:
The JewelPump (Debiotech) will be compared to the conventional pumps. Patients will treated with the JewelPump during 5 days, and with their usual pump during 5 other days.

The study will be conduct with 15 patients at the following investigation centers : Corbeil Hospital, CHU of Strasbourg, and CHRU of Marseille.

ELIGIBILITY:
Inclusion Criteria:

* Patients type 1 diabetics treated by external insulin pump;
* Patients with HbA1c < 8.5%
* Patients who signed consent

Exclusion Criteria:

* Patients type 2 diabetics
* Patients who have all serious diseases that could interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Time spent in glycemic area 70-180 mg / dl, measured continuously for 5 days with a continuous glucose monitoring (CGM) DEXCOM G4 | up to 5 days of each treatment period
  Evaluate the non-inferiority of JewelPump compared to the usual pump patient, on glycemic control.

SECONDARY OUTCOMES:
Time spent in the strict glycemic area 80-140 mg / dl | up to 5 days of each treatment period
  Evaluate the superiority of JewelPump versus usual pump;

OTHER OUTCOMES:
Time spent below 70 mg / dl | up to 5 days in each treatment period
Time spent above 180mg/dl; | up to 5 days in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia FRANC, MD, Principal Investigator — Centre Hospitalier Sud Francilien; Nathalie JEANDIDIER, Pr., Principal Investigator — University Hospital, Strasbourg, France; Denis RACCAH, Pr., Principal Investigator — Centre Hospitalier Universitaire de Marseille; Guillaume CHARPENTIER, MD, Study Chair — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète
Locations (3):
- France (3):
  - Centre Hospitalier Sud Francilien, Évry
  - CHU Marseille-Hôpital Nord, Marseille
  - CHU Strasbourg, Strasbourg